CLINICAL TRIAL: NCT02288910
Title: Blood Volume Assessment of Hepatocellular and Metastatic Carcinomas in the Liver
Status: Completed | Type: Observational
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 14030305
Record Dates: First submitted 2014-11-05; First posted 2014-11-11 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Hepatocellular Carcinoma; Metastatic Carcinoma to the Liver
Keywords: Liver Perfusion; DynaCT Perfusion; Radioembolization; Chemoembolization
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This project investigates the feasibility of assessing the relative blood volume of carcinomas in patients with Hepatocellular Carcinoma (HCC) and liver metastases from pancreatic or colorectal cancer compared to normal liver from DynaCT acquisitions on an interventional platform.

DETAILED DESCRIPTION:
This project will enroll patients with non-diffuse liver disease who are candidates for chemo or radioembolization to treat or manage the disease during an image guided intervention. Subjects will undergo a CT perfusion study of the liver prior to the radioembolizaiton mapping procedure or prior to the chemoembolization treatment. During the radioembolization mapping or chemoembolization procedure, 2 DynaCT acquisitions on the interventional C-arm will be acquired (the second during an injection of an iodinated contrast material) and will be processed using Siemens' PBV software to generate blood volume maps. The diagnostic accuracy of the two approaches to assess the vascularity of the tumors will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* HCC or metastatic liver disease
* Candidate for radioembolization or chemoembolization

Exclusion Criteria:

* Pregnant
* Iodine allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with non-diffuse hepatocellular carcinoma or metastatic liver disease
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2014-11; Primary Completion 2019-07 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of PBV maps | 1 year
  The accuracy of the DynaCT BV protocol as an indicator of healthy vs. liver tumor compared to the body CT perfusion study will evaluated using a receiver operating characteristic curve.

SECONDARY OUTCOMES:
Relationship between blood volume values and patient treatment response | 1,4,7,13,19 months
  The relationship between the BV values obtained by both methods and treatment response (as measured by RECIST values) will be evaluated by a logistic regression model
PBV blood volume value accuracy | 1 year
  A Spearman's correlation coefficient will be used to test the rank-based correlation of the BV values in tumor from the DynaCT BV acquisition to the body CT perfusion values. Furthermore, a paired t-test will be used to test for differences in BV using the two approaches.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Supanich, PH.D., Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States